CLINICAL TRIAL: NCT03438929
Title: Clinical Evaluation of Diolaze XL Blended Mode for Hair Removal
Brief Title: Evaluation of Diolaze XL Blended Mode for Hair Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO607227A
Record Dates: First submitted 2018-02-12; First posted 2018-02-20 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-02

CONDITIONS: Hair Removal
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Diode laser — Diolaze XL blended modes diode laser

SUMMARY:
The objective of this clinical study is to evaluate safety and efficiency of Diolase XL blended modes for hair removal. The handpieces tested were a blend of 755nm/810nm and 810nm/1064nm. At least 30 female subjects seeking hair removal treatment will be enrolled. Treatment sites will be o groins and axillae. Study design included 3 treatment sessions 4 weeks apart and follow-up after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult females between the ages of 18-65, seeking hair removal treatments.
* Subjects skin type II-V.
* Subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, (including the permission to use photography).
* Subjects should be willing to comply with the study procedure and schedule, including the follow up visit, to refrain from using any other aesthetic treatment methods in the treatment areas such as other hair removal methods (wax, IPL, laser), Botox or other technologies for hyperhidrosis or rejuvenation for the last 6 months and during the entire study period and to remain unshaven for a minimum of 3 days before their visit.

Exclusion Criteria:

* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes, thyroid dysfunction, polycystic ovary and hormonal virilization.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Known skin photosensitivity or using drugs increasing skin photosensitivity.
* Diseases that may be stimulated by light, such as epilepsy, lupus and urticaria.
* Six months delay is recommended if other recent treatments like light, laser or RF were performed on the same area.
* Treating over tattoo and permanent make-up.
* Fresh tan from sun, sunbeds or chemicals or planned excessive sun exposure.
* Vitiligo.
* As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-10 (Actual)

PRIMARY OUTCOMES:
Hair reduction | 3 months follow-up
  Hair reduction of at least 30% at follow-up visit comparing to baseline count.
Recording of frequency, severity and causality of adverse events (Safety) | 3 months follow-up
  Observation, assessment and recording of reactions by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Hela Goren, Ph.D., Study Director — InMode MD Ltd.
Locations (1):
- InMode MD Ltd., Yoqneam, Israel